CLINICAL TRIAL: NCT02179216
Title: Evaluation of the Effect of Hydration About Orthostatic Hypotension in the Elderly. Difference With Venous Compression. A Randomized Controlled Crossover Trial.
Brief Title: Evaluation of the Effect of Hydration About Orthostatic Hypotension in the Elderly. Difference With Venous Compression
Acronym: CHHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2014-A00695-42
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Orthostatic Hypotension
Keywords: Orthostatic hypotension in the elderly; Efficacity of Hydration; Difference between hydratation and venous contention
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydration (Active Comparator): •Group 1: First day, Orthostatic Hypotension test after hydration by three large glasses of clear liquid (33cl). Second day, Orthostatic Hypotension test with venous contention in the morning.
  Interventions: Other: Hydration; Other: Venous contention
- Venous contention (Active Comparator): •Group 2: First day, Orthostatic Hypotension test after implementation of venous contention in the morning. Second day, Orthostatic Hypotension test after hydration by three large glasses of clear liquid (33cl).
  Interventions: Other: Hydration; Other: Venous contention

INTERVENTIONS:
Other: Hydration — Hydratation the first day in the arm 1 Hydration the second day in the arm 2
Other: Venous contention — Venous contention the second day in the arm 1 Venous contention the first day in the arm 2

SUMMARY:
Primary objective: To compare the decrease in systolic blood pressure between hydration and venous contention when switching to a standing position. Hypothesis in that hydration is better than venous contention.

Secondary objective: To evaluate the effect of hydration on lowering systolic blood pressure during the passage standing in elderly patients with orthostatic hypotension.

Inclusion criteria: Patient aged over 75 years old with orthostatic hypotension proved to 1 and / or 3 min

DETAILED DESCRIPTION:
Day 0: confirmation of the orthostatic hypotension, without prevented measures

Two groups randomized :

* Group 1: First day (day 1), Orthostatic Hypotension test after hydration by three large glasses of clear liquid (33cl). Second day (day 2), Orthostatic Hypotension test with venous contention in the morning.
* Group 2: First day (day 1), Orthostatic Hypotension test after implementation of venous contention in the morning. Second day (day 2), Orthostatic Hypotension after hydration by three large glasses of clear liquid (33cl).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 and older with orthostatic hypotension proved to 1 and / or 3 minutes.
* Written consent of the subject
* Hospitalization or stay expected minimum 3 days
* Affiliation to a social security scheme

Exclusion Criteria:

* bedridden patient or without possibility of verticalization
* Patient who can't stand up (pulmonary embolism with high risk)
* Patient who refuse to participate in the study
* Patient with legal protection
* State or condition that may affect the stability of blood pressure during the study (hyperthermia, modification antihypertensive treatments less than 48 hours before inclusion...)
* Pathology preventing hydration: Heart failure with less than 1 Liter water restriction, swallowing disorders preventing hydration orally, inability to nutrition and hydration orally
* Intravenous or subcutaneous hydration (intravenous or subcutaneous treatments not included)
* Patient who can't have venous contention: Blue phlebitis, septic thrombosis, arteritis with score less than 0.6, varicose ulcers during treatment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
difference in systolic blood pressure between sitting and standing at 1 and 3 minutes between hypotension test with hydration and hypotension test with venous contention | during 3 days: day 0, day 1, day 2

SECONDARY OUTCOMES:
difference in systolic blood pressure between sitting and standing at 1 and 3 minutes between hypotension test with hydration and hypotension test without prevention | during 3 days: at day 0, day 1, day 2

CONTACTS AND LOCATIONS:
Overall Officials: Athanase Benetos, Pr, Principal Investigator — CHU Brabois
Locations (2):
- France (2):
  - Centre Hospitalier Régional Universitaire de Nancy, Nancy
  - Maison Hospitalière Saint Charles, Nancy

REFERENCES:
- [Background] Gorelik O, Almoznino-Sarafian D, Litvinov V, Alon I, Shteinshnaider M, Dotan E, Modai D, Cohen N. Seating-induced postural hypotension is common in older patients with decompensated heart failure and may be prevented by lower limb compression bandaging. Gerontology. 2009;55(2):138-44. doi: 10.1159/000141920. Epub 2008 Jun 27. PMID 18583904
- [Background] Tyberghein M, Philips JC, Krzesinski JM, Scheen AJ. [Orthostatic hypotension: definition, symptoms, assessment and pathophysiology]. Rev Med Liege. 2013 Feb;68(2):65-73. French. PMID 23469486
- [Background] Schols JM, De Groot CP, van der Cammen TJ, Olde Rikkert MG. Preventing and treating dehydration in the elderly during periods of illness and warm weather. J Nutr Health Aging. 2009 Feb;13(2):150-7. doi: 10.1007/s12603-009-0023-z. PMID 19214345
- [Background] Rutan GH, Hermanson B, Bild DE, Kittner SJ, LaBaw F, Tell GS. Orthostatic hypotension in older adults. The Cardiovascular Health Study. CHS Collaborative Research Group. Hypertension. 1992 Jun;19(6 Pt 1):508-19. doi: 10.1161/01.hyp.19.6.508. PMID 1592445